CLINICAL TRIAL: NCT04674865
Title: Effects of Anulom-Vilom Pranayama/ Alternate Nostril Breathing on Cardiorespiratory Functions in Phase 1 Post CABG Patients
Brief Title: Alternate Nostril Breathing on Cardiorespiratory Functions in Phase 1 Post CABG Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00698 Saleha Komal
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Post-cardiac Surgery
Keywords: Alternate nostril breathing; Cardiorespiratory parameters; Cardiovascular disease; Arterial blood gases; Pulmonary function test
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment protocol group (Active Comparator): Standardized treatment protocol including chest physical therapy as well as limb physical therapy and functional mobility was addressed.
  Interventions: Other: Standardized Physical therapy protocol
- ANB group (Experimental): 2 sessions per day was added to the standardized treatment protocol
  Interventions: Other: Alternate nostrils breathing

INTERVENTIONS:
Other: Standardized Physical therapy protocol — Standardized Phase 1 protocol without for 7 days without ANB sessions.
  Arms: Conventional treatment protocol group
Other: Alternate nostrils breathing — Alternate nostrils breathing 2 sessions per day
  Arms: ANB group

SUMMARY:
The aim of this study is to investigate effects of Anulom vilom pranayama/ Alternate nasal breathing (ANB) on cardio-respiratory parameters including vitals i.e. heart rate, blood pressure, chest expansion, arterial blood gases (ABGs), pulmonary function test and functional capacity in phase 1 post CABG patients. This study will help Cardiopulmonary physiotherapists to incorporate evidence based protocols for Coronary Artery Bypass Graft Surgery (CABG) in phase 1 of cardiac rehabilitation.

DETAILED DESCRIPTION:
Breathing is essential function of the body. Learning of breath regulation permits to control body's different mechanisms. "Pranayama" means control of breathing. ANB training consist of mindful breathing. Alternate nostril breathing works on regulating respiratory pattern, improvement of ventilation, clearance of lungs from retaining mucus, decrease in work of breathing and relax the mind and body. Alternate-nostril breathing (ANB) is one type of pranayama that contains inhalation from left side nostril and exhalation by right nostril afterwards inhalation by right nostril and exhalation from left nostril. This technique includes inhalation, exhalation and in advance training retention is also include. Its duration can be vary as depends on person's own capacity. ANB is usually considered to release mental conflict and stimulate mental stability and physical health. There are various studies to evaluate the outcomes of alternate breathing technique on definite functions of cognitive and physiological systems. cardiovascular disorder is the foremost reason of passing away for both gender. Coronary Artery Disease(CAD) is narrowing or obstruction of the arteries/vessels (which deliver nutrients and oxygen to the heart) as a result of atherosclerotic plaque or clot formed in the arteries. 50% patient with CAD showed their first symptoms as cardiac arrest. In western world CAD is the most common root for death. In worldwide, with the risk factors of Smoking, High cholesterol, Hypertension, Diabetes, Emotional stress, Obesity and Sedentary life, each year 3.8 million men & 3.4 million women die due to CAD. Coronary Artery Bypass Grafting(CABG) is most common surgery performed for CAD. This operation can be one week of daily training of Pranayama revealed to induce improvement in the sympathetic tone. Yoga practice along with different breathing exercises improve cardiac output, reduce hepatic, renal blood flow and increases blood flow in cerebral peripheral vessels. Heart rate vary with every single thought and environmental situation. In Anulom - Vilom pranayama, practitioner not only tries to breathe, but at the same moment, retain his focus on the action of breathing, leading to get awareness. This act of attentiveness distract him from tough concerns and evokes relax response. In this stress free state, parasympathetic nerve action supersedes sympathetic nerve's activity lead to noteworthy reduction in systolic blood pressure. Short term training of Anulom vilom pranayama indicated a substantial impact on Systolic Blood Pressure and showed an encouraging outcome on mental and digestive functions. Studies conducted showed that three months Yoga training is highly beneficial for the improvement of blood pressure and heart rate in stage 1 hypertensive patients. Role for ANB in hypertensive people is beneficial to perform focused tasks without sympathetic activation (based on an increased BP). Practice of ANB in Prehypertensive obese young adults for 15 min daily showed a significant improvement in cardiovascular parameters.

ANB plays a significant role in improving the various ventilatory functions of lungs, vital capacity and PEFR in pranayama practicing subjects. Increase in VC signifies complete emptying and fullness of air. Blood Pressure and Pulse rate is related with Cardio Vascular System, which is controlled by Autonomous nervous System (ANS). Pranayama accompanied by breath control increases cardiac output, decreases hepatic, renal blood flow and increases cerebral peripheral vessels blood flow. Heart rate varies with single thought and thoughtless condition Blood Pressure and Pulse rate is related with Cardio Vascular System, which is controlled by Autonomous nervous System (ANS). Pranayama accompanied by breath control increases cardiac output, decreases hepatic, renal blood flow and increases cerebral peripheral vessels blood flow. Heart rate varies with single thought and thoughtless condition Blood Pressure and Pulse rate is related with Cardio Vascular System, which is controlled by Autonomous nervous System (ANS). ANB accompanied by breath control increases cardiac output, decreases hepatic, renal blood flow and increases cerebral peripheral vessels blood flow. Heart rate varies with single thought and thoughtless condition Blood Pressure and Pulse rate is related with Cardio Vascular System, which is controlled by Autonomous nervous System (ANS). ANB accompanied by breath control increases cardiac output, decreases hepatic, renal blood flow and increases cerebral peripheral vessels blood flow. Heart rate varies with single thought and thoughtless condition Blood Pressure and Pulse rate is related with Cardio Vascular System, which is controlled by Autonomous nervous System (ANS). ANB accompanied by breath control increases cardiac output, decreases hepatic, renal blood flow and increases cerebral peripheral vessels blood flow. Heart rate varies with single thought and thoughtless condition The worth of physiotherapy skills used for patients after coronary artery bypass surgery (CABG) is well recognized. It is a life-saving process which is usually related with substantial postoperative pain. Various lungs functions may become compromised, or visibly vain, because of severe chest pain and there is frequently chances to develop restrictive lung disease after cardiac surgery. Though painkillers may be effective to diminish the pain but they have side effects which include respiratory depression or respiratory muscles weakness. Hence, development of chemical free approaches for effective pain control is a long standing interest. After Coronary Artery Bypass Grafting (CABG), the quality of life (QOL) is main factor to morbidity and mortality. Adding of Yoga Based Lifestyle Program (YLSP) to cardiac rehabilitation has established a valuable and actual improvement in ejection fraction and decreasing in risk factor profiles.

Many studies have been done on the efficacy of this exercise practice in healthy and clinical populations on cardiovascular and the autonomic functions. Numerous investigations have recommended that ANB improves the balance between sympathetic vagal and parasympathetic dominance. Training of ANB after CABG improves chest expansion, peak expiratory flow rate and decrease in pain. ANB along with conventional physiotherapy play a key role in improving Respiratory function and depression issues in CABG patients.

Literature reviewed from different search engines has shown that alternate breathing technique has significant positive effects on cardiorespiratory functions but very little literature has been found specifically on phase 1 post CABG studies, regarding to ANB effect.

ELIGIBILITY:
Inclusion Criteria:

- Patient's undergoing CABG surgery.

Exclusion Criteria:

* With any difficulty in communication.
* Unstable vital signs
* Those who are smokers.
* Other severe complications like diabetes, stroke or cancer.
* Patient with any respiratory / other pathologies will not be included

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow rate (PEFR) | 7 days
  Peak expiratory flow rate (PEFR) measured through digital spirometer. Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings.
Forced vital capacity (FVC) | 7 days
  Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal.
Forced expiratory volume in 1sec (FEV1) | 7 days
  Forced expiratory volume in 1sec (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal.
FVC/FEV1 | 7 days
  FVC/FEV1 measured through digital spirometer. The normal value for the FEV1/FVC ratio is 70% (and 65% in persons older than age 65).
Arterial Blood Gases | 7 days
  An arterial blood gas (ABG) test measures oxygen and carbon dioxide levels in the blood. It also measures body's acid-base (pH) level, which is usually in balance when a person is healthy.

SECONDARY OUTCOMES:
Chest expansion | 7 days
  Chest expansion at xiphoid level measured by finding the difference in measurements during inhalation and exhalation.
Heart rate | 7 days
  Heart rate is measured as part of vitals through heart rate monitor.
Systolic and diastolic blood pressure | 7 days
  Blood pressure is measured through sphygmomanometer
Oxygen Saturation (SPO2) | 7 days
  Oxygen saturation measured through pulse oximeter as part of vitals
Six Minute Walk Test (6MWT) | 7 days
  6MWT is used to assess the functional capacity of patients by calculating the distance covered in a time period of 6 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Rawalpindi, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Shakouri SK, Salekzamani Y, Taghizadieh A, Sabbagh-Jadid H, Soleymani J, Sahebi L, Sahebi R. Effect of respiratory rehabilitation before open cardiac surgery on respiratory function: a randomized clinical trial. J Cardiovasc Thorac Res. 2015;7(1):13-7. doi: 10.15171/jcvtr.2015.03. Epub 2015 Mar 29. PMID 25859310
- [Background] Raghuram N, Parachuri VR, Swarnagowri MV, Babu S, Chaku R, Kulkarni R, Bhuyan B, Bhargav H, Nagendra HR. Yoga based cardiac rehabilitation after coronary artery bypass surgery: one-year results on LVEF, lipid profile and psychological states--a randomized controlled study. Indian Heart J. 2014 Sep-Oct;66(5):490-502. doi: 10.1016/j.ihj.2014.08.007. Epub 2014 Aug 28. PMID 25443601
- [Background] Kamath A, Urval RP, Shenoy AK. Effect of Alternate Nostril Breathing Exercise on Experimentally Induced Anxiety in Healthy Volunteers Using the Simulated Public Speaking Model: A Randomized Controlled Pilot Study. Biomed Res Int. 2017;2017:2450670. doi: 10.1155/2017/2450670. Epub 2017 Oct 11. PMID 29159176
- [Background] Saoji AA, Raghavendra BR, Manjunath NK. Effects of yogic breath regulation: A narrative review of scientific evidence. J Ayurveda Integr Med. 2019 Jan-Mar;10(1):50-58. doi: 10.1016/j.jaim.2017.07.008. Epub 2018 Feb 1. PMID 29395894
- [Background] Zou Y, Zhao X, Hou YY, Liu T, Wu Q, Huang YH, Wang XH. Meta-Analysis of Effects of Voluntary Slow Breathing Exercises for Control of Heart Rate and Blood Pressure in Patients With Cardiovascular Diseases. Am J Cardiol. 2017 Jul 1;120(1):148-153. doi: 10.1016/j.amjcard.2017.03.247. Epub 2017 Apr 12. PMID 28502461